CLINICAL TRIAL: NCT01877915
Title: A Randomized, Double-blind, Event-driven, Multicenter Study Comparing the Efficacy and Safety of Rivaroxaban With Placebo for Reducing the Risk of Death, Myocardial Infarction or Stroke in Subjects With Heart Failure and Significant Coronary Artery Disease Following an Episode of Decompensated Heart Failure
Brief Title: A Study to Assess the Effectiveness and Safety of Rivaroxaban in Reducing the Risk of Death, Myocardial Infarction or Stroke in Participants With Heart Failure and Coronary Artery Disease Following an Episode of Decompensated Heart Failure
Acronym: COMMANDER HF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR101940; RIVAROXHFA3001 (Other: Janssen Research & Development, LLC); 2013-000046-19 (EudraCT Number)
Record Dates: First submitted 2013-06-12; First posted 2013-06-14 (Estimated); Results first posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-04

CONDITIONS: Heart Failure; Coronary Artery Disease
Keywords: Heart Failure; Coronary Artery Disease; Stroke; Myocardial Infarction; Anticoagulation
MeSH Terms: conditions — Heart Failure; Coronary Artery Disease; Stroke; Myocardial Infarction | interventions — Rivaroxaban; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rivaroxaban 2.5 mg (Experimental): Each participant will receive 2.5 mg of rivaroxaban twice daily with standard of care for heart failure and coronary artery disease (as prescribed by the participant's managing physician).
  Interventions: Drug: Rivaroxaban; Other: Standard of care for heart failure and coronary artery disease
- Placebo (Placebo Comparator): Each participant will receive matching placebo twice daily with standard of care for heart failure and coronary artery disease (as prescribed by the participant's managing physician).
  Interventions: Drug: Placebo; Other: Standard of care for heart failure and coronary artery disease

INTERVENTIONS:
Drug: Rivaroxaban — Each participant, randomly allocated to the rivaroxaban arm, will receive one 2.5 mg tablet of rivaroxaban orally (by mouth) twice daily (once in the morning and once in the evening at approximately the same time each day) until the global treatment end date (GTED) (defined as the date when 1200 primary efficacy outcome events have occurred). Rivaroxaban will be given with standard of care for heart failure and coronary artery disease (as prescribed by the participant's managing physician).
  Arms: Rivaroxaban 2.5 mg
Drug: Placebo — Each participant, randomly allocated to the placebo arm, will receive one matching placebo tablet orally twice daily (once in the morning and once in the evening at approximately the same time each day) until the GTED. Placebo will be given with standard of care for heart failure and coronary artery disease (as prescribed by the participant's managing physician).
  Arms: Placebo
Other: Standard of care for heart failure and coronary artery disease — Each participant's standard of care for heart failure and coronary artery disease (as prescribed by the participant's managing physician) should be continued throughout the study.

SUMMARY:
The purpose of this study is to assess the effectiveness and safety of rivaroxaban compared with placebo (inactive medication), in reducing the risk of death, myocardial infarction or stroke in participants with heart failure and significant coronary artery disease following an episode of decompensated heart failure.

DETAILED DESCRIPTION:
This is a randomized (the study medication is assigned by chance), double-blind (neither physician nor participant knows the identity of the assigned treatment), parallel group (each participant group receives different treatments simultaneously), event driven (the study duration is determined by the time taken for a specific number of events to occur), multicenter study to assess the effectiveness and safety of rivaroxaban compared with placebo, in reducing the risk of death, myocardial infarction or stroke in participants with heart failure and significant coronary artery disease following an episode of decompensated heart failure. Participants will be randomly assigned in a 1:1 ratio to receive either rivaroxaban or placebo (each in addition to standard of care for heart failure and coronary artery disease as prescribed by their managing physician). The study will consist of a screening phase, a double-blind treatment phase, and a follow-up after the sponsor-announced global treatment end date (GTED, defined as the date when 1200 primary efficacy outcome events are predicted to have occurred). The double-blind treatment phase is estimated to last for 6 to 54 months. Participants will discontinue study drug after taking both their morning and evening doses on the GTED and will return to the study center for the end-of-study visit (between 15 and 45 days but no sooner than 15 days after the GTED). Patient safety will be monitored throughout the study. The average study duration for participants is expected to be approximately 29 months. The study drug, rivaroxaban, is approved in the United States and in multiple countries around the world for the prevention and treatment of a number of thrombosis-mediated conditions.

ELIGIBILITY:
Inclusion Criteria:

* Must have symptomatic heart failure for at least 3 months prior to Screening
* Participants must have an episode of decompensated heart failure (index event) requiring (a) an overnight stay [that is, staying past midnight] in a hospital, emergency department, or medical facility with the capability of treating with intravenous medications and observing heart failure patients before randomization or (b) an unscheduled outpatient visit to a heart failure management center, where parenteral therapy is required for heart failure stabilization. An episode of decompensated heart failure is defined as symptoms of worsening dyspnea or fatigue, objective signs of congestion such as peripheral edema or ascites, and/or adjustment of pre-hospitalization/outpatient visit heart failure medications. Participants are eligible for randomization at discharge from the facility treating the index event and up to 30 days after discharge if they are in stable condition
* Must have a documented left ventricular ejection fraction (LVEF) of less than or equal to 40 percent (%) within 1 year before randomization
* Must have evidence of significant coronary artery disease
* Must be medically stable in terms of their heart failure clinical status at the time of randomization
* Must have a brain natriuretic peptide (BNP) level greater than or equal to (>=) 200 picogram per milliliter (pg/mL) or N-terminal-proBNP (NT-proBNP) level >=800 pg/mL (preferred assay) during the Screening period and before randomization

Exclusion Criteria:

* Any condition that, in the opinion of the investigator, contraindicates anticoagulant therapy or would have an unacceptable risk of bleeding, such as, but not limited to, active internal bleeding, clinically significant bleeding, bleeding at a noncompressible site, or bleeding diathesis within 28 days of randomization
* Severe concomitant disease such as (a) atrial fibrillation (AFib) or another condition that requires chronic anticoagulation (participants with isolated transient AFib may be allowed at the discretion of the treating physician investigator) and (b) Documented acute myocardial infarction (MI) during index event
* Prior stroke within 90 days of randomization
* Has been hospitalized for longer than 21 days during the index event
* Planned intermittent outpatient treatment with positive inotropic drugs administered intravenously

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5081 (Actual)
Dates: Start 2013-09-10 (Actual); Primary Completion 2018-04-19 (Actual); Study Completion 2018-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (563):
- United States (115):
  - Alexander City, Alabama
  - Birmingham, Alabama
  - Mobile, Alabama
  - Anchorage, Alaska
  - Tucson, Arizona
  - Jonesboro, Arkansas
  - Beverly Hills, California
  - Chula Vista, California
  - El Cajon, California
  - Glendale, California
  - La Mesa, California
  - Los Angeles, California
  - Newport Beach, California
  - Orange, California
  - Stockton, California
  - Torrance, California
  - Aurora, Colorado
  - Denver, Colorado
  - New Haven, Connecticut
  - Atlantis, Florida
  - Daytona Beach, Florida
  - Jupiter, Florida
  - Orlando, Florida
  - St. Petersburg, Florida
  - Tallahassee, Florida
  - Wellington, Florida
  - Winter Haven, Florida
  - Athens, Georgia
  - Atlanta, Georgia
  - Cumming, Georgia
  - Macon, Georgia
  - Tucker, Georgia
  - Chicago, Illinois
  - Evanston, Illinois
  - Fairview Heights, Illinois
  - Peoria, Illinois
  - Rockford, Illinois
  - Urbana, Illinois
  - Anderson, Indiana
  - Indianapolis, Indiana
  - Merrillville, Indiana
  - Munster, Indiana
  - South Bend, Indiana
  - Iowa City, Iowa
  - Elizabethtown, Kentucky
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Owensboro, Kentucky
  - Bossier City, Louisiana
  - Hammond, Louisiana
  - Shreveport, Louisiana
  - Slidell, Louisiana
  - Biddeford, Maine
  - Baltimore, Maryland
  - Columbia, Maryland
  - Randallstown, Maryland
  - Bay City, Michigan
  - Grand Blanc, Michigan
  - Mount Clemens, Michigan
  - Pontiac, Michigan
  - Ypsilanti, Michigan
  - Saint Paul, Minnesota
  - Springfield, Missouri
  - St Louis, Missouri
  - Washington, Missouri
  - Lincoln, Nebraska
  - Las Vegas, Nevada
  - Bridgewater, New Jersey
  - Elmer, New Jersey
  - Haddon Heights, New Jersey
  - Manalapan, New Jersey
  - Ridgewood, New Jersey
  - Sewell, New Jersey
  - Albuquerque, New Mexico
  - Buffalo, New York
  - Cortlandt Manor, New York
  - Jamaica, New York
  - Mineola, New York
  - New York, New York
  - Charlotte, North Carolina
  - High Point, North Carolina
  - Pinehurst, North Carolina
  - Canton, Ohio
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Fairfield, Ohio
  - Kettering, Ohio
  - Bartlesville, Oklahoma
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Doylestown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Sayre, Pennsylvania
  - Sellersville, Pennsylvania
  - Wynnewood, Pennsylvania
  - Yardley, Pennsylvania
  - York, Pennsylvania
  - Charleston, South Carolina
  - Sioux Falls, South Dakota
  - Nashville, Tennessee
  - Cypress, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Huntsville, Texas
  - Kingwood, Texas
  - Lubbock, Texas
  - McKinney, Texas
  - Burlington, Vermont
  - Newport News, Virginia
  - Bellingham, Washington
  - Tacoma, Washington
  - Huntington, West Virginia
- Argentina (16):
  - Bahía Blanca
  - Buenos Aires
  - Caba
  - Córdoba
  - La Plata
  - Mar del Plata
  - Mendoza
  - Merlo
  - Quilmes
  - Resistencia
  - Rosario
  - San Miguel de Tucumán
  - San Nicolás
  - Santa Fe
  - Santiago del Estero
  - Vicente López
- Australia (10):
  - Bedford
  - Cairns
  - Concord
  - Darlinghurst
  - Hobart
  - Launceston
  - Perth
  - Sydney
  - Wollongong
  - Woolloongabba
- Brazil (23):
  - Belém
  - Belo Horizonte
  - Blumenal
  - Brasília
  - Campina Grande do Sul
  - Campinas
  - Campo Grande
  - Canoas
  - Curitiba
  - Goiânia
  - Marília
  - Passo Fundo
  - Porto Alegre
  - Recife
  - Ribeirão Preto
  - Rio de Janeiro
  - Salvador
  - São Jose Do Rio Preto
  - São Paulo
  - São Pedro
  - Tatuí
  - Uberlândia
  - Votuporanga
- Bulgaria (12):
  - Blagoevgrad
  - Burgas
  - Dimitrovgrad
  - Kazanlak
  - Pazardzhik
  - Pleven
  - Plovdiv
  - Rousse
  - Sofia
  - Stara Zagora
  - Varna
  - Veliko Tarnovo
- Canada (11):
  - Edmonton, Alberta
  - Maple Ridge, British Columbia
  - St. John's, Newfoundland and Labrador
  - Halifax, Nova Scotia
  - Cambridge, Ontario
  - Kitchener, Ontario
  - London, Ontario
  - Ottawa, Ontario
  - Scarborough Village, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- China (27):
  - Baotou
  - Beijing
  - Changchun
  - Changsha
  - Chengdu
  - Daqing
  - Guangzhou
  - Haikou
  - Hangzhou
  - Hunan
  - Jinan
  - Jining
  - Lanzhou
  - Nanchang
  - Nanjing
  - Nanning
  - Qingdao
  - Shanghai
  - Shenyang
  - Shijiazhuang
  - Suzhou
  - Taiyuan
  - Tianjin
  - Wuhan
  - Xi'an
  - Yangzhou
  - Yichang
- Czechia (17):
  - Brno
  - Hodonín
  - Hradec Králové
  - Hranice
  - Karlovy Vary
  - Kladno
  - Kolín
  - Litomyšl
  - Mladá Boleslav
  - Olomouc
  - Plze?-Bory
  - Prague
  - Praha 8 - Libe?
  - Slaný
  - Teplice
  - Uherské Hradišt?
  - Valašské Mezi?í?í
- Denmark (5):
  - Esbjerg
  - Herlev
  - Hjørring
  - Hvidovre
  - Køge
- Tallinn, Estonia
- France (12):
  - Besançon
  - Bron
  - Chambray-lès-Tours
  - Corbeil-Essonnes
  - Lille
  - Montpellier
  - Nantes
  - Nice
  - Pau
  - Rouen
  - Toulouse
  - Vandœuvre-lès-Nancy
- Germany (19):
  - Berlin
  - Bielefeld
  - Bonn
  - Coburg
  - Dresden
  - Halle
  - Hamburg
  - Heidelberg
  - Konstanz
  - Langen
  - Leipzig
  - Ludwigshafen
  - Magdeburg
  - Mainz
  - Markkleeberg
  - Papenburg
  - Stuttgart
  - Ulm
  - Witten
- Greece (5):
  - Athens
  - Heraklion -Crete
  - Larissa
  - Thessalonikis
  - Voula
- Hungary (10):
  - Balatonfüred
  - Berettyóújfalu
  - Budapest
  - Győr
  - Miskolc
  - Nagykanizsa
  - Szekszárd
  - Székesfehérvár
  - Szolnok
  - Zalaegerszeg
- Japan (51):
  - Aichi
  - Chiba
  - Chikushino-shi
  - Ehime
  - Fukuoka
  - Gifu
  - Gunma
  - Hatsukaichi
  - Hitachi
  - Hokkaido
  - Hyōgo
  - Ibaraki
  - Ishikawa
  - Izumo
  - Kagawa
  - Kahoku-District
  - Kanagawa
  - Kobe
  - Komatsushima-shi
  - Koshigaya-shi
  - Kumamoto
  - Kyoto
  - Miyazaki
  - Nagano
  - Nagasaki
  - Nagoya
  - Niigata
  - Okayama
  - Okinawa
  - Osaka
  - Ōita
  - Saga
  - Saitama
  - Sapporo
  - Sendai
  - Shiga
  - Shimane
  - Shizuoka
  - Tachikawa
  - Takaraduka
  - Tochigi
  - Tokushima
  - Tokyo
  - Toyama
  - Toyoake
  - Tsu
  - Wakayama
  - Yamaguchi
  - Yatsushiro
  - Yokohama
  - Yonago
- Latvia (6):
  - Daugavpils
  - Kuldīga
  - Liepāja
  - Riga
  - Sigulda
  - Ventspils
- Lithuania (6):
  - Alytus
  - Kaunas
  - Klaipėda
  - Panevezys
  - Šiauliai
  - Vilnius
- Malaysia (8):
  - Cheras
  - George Town
  - Johor Bahru
  - Kota Kinabalu
  - Kuala Lumpur
  - Kuala Selangor
  - Kuching
  - Selayang Baru Utara
- Mexico (16):
  - Aguascalientes
  - Benito Juárez
  - Chihuahua City
  - Culiacán
  - Durango
  - Guadalajara
  - León
  - Mexico City
  - México
  - Oaxaca City
  - Pachuca
  - Puebla City
  - Querétaro
  - San Luis Potosí City
  - Tampico
  - Veracruz
- Netherlands (13):
  - Almere Stad
  - Amsterdam
  - Blaricum
  - Breda
  - Deventer
  - Doetinchem
  - Ede
  - Groningen
  - Heerlen
  - Helmond
  - Maastricht
  - Meppel
  - Tilburg
- Poland (30):
  - Będzin
  - Gdynia
  - Gliwice
  - Grodzisk Mazowiecki
  - Inowrocław
  - Katowice
  - Kielce
  - Krakow
  - Kutno
  - Lodz
  - Lubin
  - Lublin
  - Myślenice
  - Olsztyn
  - Ostrowiec Świętokrzyski
  - Ostrołęka
  - Oświęcim
  - Puławy
  - Płock
  - Rabka-Zdrój
  - Skierniewice
  - Starogard Gdański
  - Szczecin
  - Torun
  - Warsaw
  - Wroclaw
  - Włocławek
  - Zabrze
  - Zamość
  - Łódż
- Portugal (11):
  - Almada
  - Aveiro
  - Braga
  - Carnaxide
  - Coimbra
  - Covilha
  - Leiria
  - Lisbon
  - Matosinhos Municipality
  - Viana do Castelo
  - Vila Real
- Romania (16):
  - Bacau
  - Baia Mare
  - Brasov
  - Brăila
  - Bucharest
  - Buzău
  - Cluj-Napoca
  - Craiova
  - Focşani
  - Galati
  - Iași
  - Oradea
  - Piteşti
  - Sibiu
  - Târgu Mureş
  - Timișoara
- Russia (27):
  - Arkhangelsk
  - Barnaul
  - Chita
  - Ivanovo
  - Izhevsk
  - Kaluga
  - Kemerovo
  - Kirov
  - Krasnoyarsk
  - Kursk
  - Moscow
  - Moscow, Zelenograd
  - Nizhny Novgorod
  - Novosibirsk
  - Orenburg
  - Perm
  - Rostov-on-Don
  - Ryazan
  - Saint Petersburg
  - Samara
  - Saratov
  - Syktyvkar
  - Tomsk
  - Tyumen
  - Voronezh
  - Yaroslavl
  - Yekaterinburg
- Slovakia (8):
  - Banská Bystrica
  - Bardejov
  - Košice
  - Lučenec
  - Moldava nad Bodvou
  - Nitra
  - Považská Bystrica
  - Svidník
- South Africa (7):
  - Bloemfontein
  - Cape Town
  - Centurion
  - Durban
  - Pinelands
  - Pretoria
  - Tongaat
- South Korea (8):
  - Busan
  - Cheongju-si
  - Daegu
  - Daejeon
  - Gwangju
  - Seongnam-si
  - Seoul
  - Wŏnju
- Spain (26):
  - A Coruña
  - Alicante
  - Almería
  - Ávila
  - Barcelona
  - Burgos
  - Cáceres
  - Elche
  - Granada
  - Lorca
  - Madrid
  - Majadahonda
  - Murcia
  - Olot
  - Orihuela
  - Palma de Mallorca
  - San Juan
  - Sanlúcar de Barrameda
  - Sant Joan Despí
  - Santander
  - Seville
  - Terrassa
  - Torrevieja
  - Valencia
  - Vigo
  - Viladecans
- Sweden (5):
  - Falun
  - Jönköping
  - Ljungby
  - Stockholm
  - Uppsala
- Turkey (Türkiye) (11):
  - Ankara
  - Bursa
  - Diyarbakır
  - Eskişehir
  - Istanbul
  - Kahramanmaraş
  - Kocaeli
  - Konya
  - Kırıkkale
  - Mersin
  - Sivas
- Ukraine (16):
  - Cherkassy
  - Cherkasy
  - Dnipro
  - Donetsk
  - Kharkiv
  - Kyiv
  - Lutsk
  - Lviv
  - Odesa
  - Poltava
  - Sumy
  - Vinnitsa
  - Vinnytsia
  - Zaporizhzhia
  - Zaporizhzhya
  - Zhytomyr
- United Kingdom (15):
  - Aberdeen
  - Airdrie
  - Birmingham
  - Chesterfield
  - Chichester
  - Clydebank
  - Cottingham
  - Dudley
  - Dundee
  - East Kilbride
  - Exeter
  - Inverness
  - Manchester
  - Metropolitan Borough of Wirral
  - TA1 5DA

REFERENCES:
- [Derived] Sharma A, Caldeira D, Razaghizad A, Pinto FJ, van Veldhuisen DJ, Mehra MR, Lam CSP, Cleland J, Anker SD, Greenberg B, Ferreira JP, Zannad F. Cardiovascular effects of rivaroxaban in heart failure patients with sinus rhythm and coronary disease with and without diabetes: a retrospective international cohort study from COMMANDER-HF. BMJ Open. 2023 Aug 11;13(8):e068865. doi: 10.1136/bmjopen-2022-068865. PMID 37567750
- [Derived] Ferreira JP, Cleland JG, Lam CSP, Anker SD, Mehra MR, van Veldhuisen DJ, Byra WM, La Police DA, Pitt B, Greenberg B, Zannad F. Heart failure re-hospitalizations and subsequent fatal events in coronary artery disease: insights from COMMANDER-HF, EPHESUS, and EXAMINE. Clin Res Cardiol. 2021 Oct;110(10):1554-1563. doi: 10.1007/s00392-021-01830-1. Epub 2021 Mar 8. PMID 33686472
- [Derived] Ferreira JP, Cleland JGF, Lam CSP, van Veldhuisen DJ, Byra WM, La Police DA, Anker SD, Mehra MR, Leroy C, Eschwege V, Toussaint-Hacquard M, Rossignol P, Greenberg B, Zannad F. Impact of Geographic Region on the COMMANDER-HF Trial. JACC Heart Fail. 2021 Mar;9(3):201-211. doi: 10.1016/j.jchf.2020.11.007. Epub 2021 Feb 3. PMID 33549557
- [Derived] Cunningham JW, Ferreira JP, Deng H, Anker SD, Byra WM, Cleland JGF, Gheorghiade M, Lam CSP, La Police D, Mehra MR, Neaton JD, Spiro TE, van Veldhuisen DJ, Greenberg B, Zannad F. Natriuretic Peptide-Based Inclusion Criteria in a Heart Failure Clinical Trial: Insights From COMMANDER HF. JACC Heart Fail. 2020 May;8(5):359-368. doi: 10.1016/j.jchf.2019.12.009. Epub 2020 Mar 11. PMID 32171760
- [Derived] Mehra MR, Vaduganathan M, Fu M, Ferreira JP, Anker SD, Cleland JGF, Lam CSP, van Veldhuisen DJ, Byra WM, Spiro TE, Deng H, Zannad F, Greenberg B. A comprehensive analysis of the effects of rivaroxaban on stroke or transient ischaemic attack in patients with heart failure, coronary artery disease, and sinus rhythm: the COMMANDER HF trial. Eur Heart J. 2019 Nov 21;40(44):3593-3602. doi: 10.1093/eurheartj/ehz427. PMID 31461239
- [Derived] Greenberg B, Neaton JD, Anker SD, Byra WM, Cleland JGF, Deng H, Fu M, La Police DA, Lam CSP, Mehra MR, Nessel CC, Spiro TE, van Veldhuisen DJ, Vanden Boom CM, Zannad F. Association of Rivaroxaban With Thromboembolic Events in Patients With Heart Failure, Coronary Disease, and Sinus Rhythm: A Post Hoc Analysis of the COMMANDER HF Trial. JAMA Cardiol. 2019 Jun 1;4(6):515-523. doi: 10.1001/jamacardio.2019.1049. PMID 31017637
- [Derived] Zannad F, Anker SD, Byra WM, Cleland JGF, Fu M, Gheorghiade M, Lam CSP, Mehra MR, Neaton JD, Nessel CC, Spiro TE, van Veldhuisen DJ, Greenberg B; COMMANDER HF Investigators. Rivaroxaban in Patients with Heart Failure, Sinus Rhythm, and Coronary Disease. N Engl J Med. 2018 Oct 4;379(14):1332-1342. doi: 10.1056/NEJMoa1808848. Epub 2018 Aug 27. PMID 30146935

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 3 participants randomized twice were only counted once in the ITT analysis set (comprised of 5,022 participants).
Groups:
- Rivaroxaban: Participants received 2.5 milligram (mg) tablet of rivaroxaban orally twice daily with standard of care for heart failure and coronary artery disease (as prescribed by the participant's managing physician).
- Placebo: Participants received matching placebo orally twice daily with standard of care for heart failure and coronary artery disease (as prescribed by the participant's managing physician).
Period: Overall Study
Arm/Group | Rivaroxaban | Placebo
Started | 2507 | 2515
Completed | 2453 | 2447
Not Completed | 54 | 68
Not completed — Lost to Follow-up | 10 | 9
Not completed — Withdrawal by Subject | 42 | 55
Not completed — Other | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban | Placebo | Total
Number analyzed (Participants) | 2507 | 2515 | 5022
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (10.07) | 66.3 (10.27) | 66.4 (10.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 551 | 599 | 1150
  Male | 1956 | 1916 | 3872
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 309 | 300 | 609
  Not Hispanic or Latino | 2186 | 2203 | 4389
  Unknown or Not Reported | 12 | 12 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 10 | 21
  Asian | 362 | 365 | 727
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 29 | 36 | 65
  White | 2063 | 2065 | 4128
  More than one race | 4 | 5 | 9
  Unknown or Not Reported | 36 | 34 | 70
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 362 | 365 | 727
  Black or African American | 29 | 36 | 65
  Other | 59 | 56 | 115
  White Hispanic or Latino | 258 | 251 | 509
  White Non-Hispanic | 1799 | 1807 | 3606
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 76 | 76 | 152
  AUSTRALIA | 7 | 7 | 14
  BRAZIL | 80 | 80 | 160
  BULGARIA | 314 | 314 | 628
  CANADA | 14 | 14 | 28
  CHINA | 186 | 186 | 372
  CZECH REPUBLIC | 35 | 34 | 69
  DENMARK | 9 | 9 | 18
  FRANCE | 10 | 10 | 20
  GERMANY | 32 | 32 | 64
  GREECE | 8 | 8 | 16
  HUNGARY | 69 | 69 | 138
  ITALY | 35 | 36 | 71
  JAPAN | 133 | 132 | 265
  LATVIA | 12 | 13 | 25
  LITHUANIA | 17 | 18 | 35
  MALAYSIA | 17 | 17 | 34
  MEXICO | 73 | 73 | 146
  NETHERLANDS | 1 | 2 | 3
  POLAND | 288 | 290 | 578
  PORTUGAL | 20 | 22 | 42
  ROMANIA | 200 | 198 | 398
  RUSSIAN FEDERATION | 274 | 276 | 550
  SLOVAKIA | 41 | 41 | 82
  SOUTH AFRICA | 8 | 8 | 16
  SOUTH KOREA | 24 | 24 | 48
  SPAIN | 89 | 89 | 178
  SWEDEN | 2 | 3 | 5
  TURKEY | 96 | 96 | 192
  UKRAINE | 264 | 265 | 529
  UNITED KINGDOM | 13 | 12 | 25
  UNITED STATES | 60 | 61 | 121

OUTCOME MEASURES:

1. Primary Outcome: Event Rate of All-Cause Mortality, Myocardial Infarction (MI), or Stroke
Description: Event Rate of all-cause mortality (ACM), MI, or stroke were assessed. Event rate estimated based on the time to the first occurrence of the event were reported in the study. Event Rate / (100 patient [pt]-year [yr]) = 100*n/(total risk exposure), where n is the number of events.
Time Frame: Up to Global treatment end date (approximately 54 months)
Population: Intent-to-Treat analysis set included all randomized unique participants who signed a valid informed consent. Participants were analyzed according to the treatment group assigned, irrespective of the actual treatment received.
Measure: Number; unit: Event rate per 100 patient-year
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 2507 | 2515
Event rate per 100 patient-year | 13.44 | 14.27
Statistical Analysis 1: Comparison: Rivaroxaban vs Placebo; Statistical Analysis 1; Test type: Superiority; p = 0.270, Log Rank; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.84 to 1.05]

2. Secondary Outcome: Event Rate of Cardio Vascular Death or Re-Hospitalization for Worsening of Heart Failure (RHHF)
Description: Event rate of cardio vascular (CV) death or re-hospitalization for worsening of heart failure were assessed. Event rate estimated based on the time to the first occurrence of the event were reported in the study. Event Rate / (100 pt-yr) = 100*n/(total risk exposure), where n is the number of events.
Time Frame: Up to Global treatment end date (approximately 54 months)
Population: as for outcome 1
Measure: Number; unit: Event rate per 100 patient-year
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 2507 | 2515
Event rate per 100 patient-year | 23.32 | 23.46

3. Secondary Outcome: Event Rate of Cardio Vascular Death
Description: Event rate of cardio vascular death were assessed. CV death included deaths due to spontaneous bleeding, MI, stroke, worsening HF and arrhythmias, death due to CV procedures and sudden death. Event rate estimated based on the time to the first occurrence of the event were reported in the study. Event Rate / (100 pt-yr) = 100*n/(total risk exposure), where n is the number of events.
Time Frame: Up to Global treatment end date (approximately 54 months)
Population: as for outcome 1
Measure: Number; unit: Event rate per 100 patient-year
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 2507 | 2515
Event rate per 100 patient-year | 9.46 | 9.96

4. Secondary Outcome: Event Rate of Re-Hospitalization for Worsening of Heart Failure
Description: Event rate of re-hospitalization for worsening of heart failure were assessed. Event rate estimated based on the time to the first occurrence of the event were reported in the study. Event Rate / (100 pt-yr) = 100*n/(total risk exposure), where n is the number of events.
Time Frame: Up to Global treatment end date (approximately 54 months)
Population: as for outcome 1
Measure: Number; unit: Event rate per 100 patient-year
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 2507 | 2515
Event rate per 100 patient-year | 17.24 | 17.45

5. Secondary Outcome: Event Rate of Re-Hospitalization for Cardio Vascular Events (RHCV)
Description: Event rate due to cardio vascular events were assessed. Hospitalization for a CV Event required that participants be hospitalized (in-patient or emergency department) for greater than 24 hours and must have met the following criterion:Discharge summary with primary reason for admission listed as CV in nature (example, bleeding, arrhythmia, ACS, MI) other than HF which was captured in the HF re-hospitalization. Event rate estimated based on the time to the first occurrence of the event were reported in the study. Event Rate / (100 pt-yr) = 100*n/(total risk exposure), where n is the number of events.
Time Frame: Up to Global treatment end date (approximately 54 months)
Population: as for outcome 1
Measure: Number; unit: Event rate per 100 patient-year
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 2507 | 2515
Event rate per 100 patient-year | 13.30 | 14.04

6. Secondary Outcome: Event Rate of All-Cause Mortality (ACM) or Re-Hospitalization for Worsening Heart Failure
Description: Event rate of all-Cause Mortality (ACM) or re-Hospitalization for worsening heart failure were assessed. Event rate estimated based on the time to the first occurrence of the event were reported in the study. Event Rate / (100 pt-yr) = 100*n/(total risk exposure), where n is the number of events.
Time Frame: Up to Global treatment end date (approximately 54 months)
Population: as for outcome 1
Measure: Number; unit: Event rate per 100 patient-year
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 2507 | 2515
Event rate per 100 patient-year | 24.84 | 24.57

7. Primary Outcome: Event Rate of Either Fatal Bleeding or Bleeding Into a Critical Space With Potential for Permanent Disability
Description: Event rate of either fatal bleeding or bleeding into critical space with potential for permanent disability were assessed. Fatal bleeding event was death within 7 days after a bleeding event which required hospitalization or met International Society on Thrombosis and Haemostasis(ISTH) major bleeding definition criteria. Fatal bleeding events included those met criteria in 3 categories: 1: Any ISTH major bleeding event consider primary cause of death by investigator; 2: Any ISTH major bleeding event not considered to be primary cause of death by investigator but resulted in death within 7 days;3: Any bleeding event resulted in hospital stay and death within 7 days. Bleeding into critical space with potential for permanent disability included 7 critical spaces: intracranial, intraspinal, intraocular. Event rate estimated based on time to first occurrence of event were reported in the study. Event Rate / (100 pt-yr) = 100*n/(total risk exposure), where n is the number of events.
Time Frame: Up to 227 Weeks
Population: Safety Analysis Set included all intent-to-treat participants who received at least one dose of study drug. Here 'N' signifies number of participants who were evaluable for this outcome measure.
Measure: Number; unit: Event rate per 100 patient-year
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 2499 | 2509
Event rate per 100 patient-year
  Fatal Bleeding | 0.22 | 0.22
  Critical Space Bleeding with Permanent Disability | 0.32 | 0.48
Statistical Analysis 1: Comparison: Rivaroxaban vs Placebo; Statistical Analysis 1 (Fatal Bleeding); Test type: Superiority; p = 0.951, Log Rank; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.41 to 2.59]
Statistical Analysis 2: Comparison: Rivaroxaban vs Placebo; Statistical Analysis 2 (Bleeding in Critical Space with Potential for Permanent Disability); Test type: Superiority; p = 0.253, Log Rank; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.33 to 1.34]

8. Secondary Outcome: Event Rate of Bleeding Events That Requiring Hospitalization
Description: Event rate of bleeding events and required Hospitalization were assessed. Event rate estimated based on the time to the first occurrence of the event were reported in the study. Event Rate / (100 pt-yr) = 100*n/(total risk exposure), where n is the number of events.
Time Frame: Up to 227 Weeks
Population: as for outcome 7
Measure: Number; unit: Event rate per 100 patient-year
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 2499 | 2509
Event rate per 100 patient-year | 1.52 | 1.16

9. Secondary Outcome: Event Rate of International Society on Thrombosis and Haemostasis (ISTH) Major Bleeding Event
Description: Event rate of ISTH major bleeding event were assessed. Event rate estimated based on the time to the first occurrence of the event were reported in the study. Event Rate / (100 pt-yr) = 100*n/(total risk exposure), where n is the number of events.
Time Frame: Up to 227 Weeks
Population: as for outcome 7
Measure: Number; unit: Event rate per 100 patient-year
Arm/Group | Rivaroxaban | Placebo
Number analyzed (Participants) | 2499 | 2509
Event rate per 100 patient-year | 2.04 | 1.21

ADVERSE EVENTS:
Time Frame: Up to 54 Months
Arm/Group | Rivaroxaban | Placebo
All-Cause Mortality (participants affected / at risk) | 565/2507 | 571/2515
Serious Adverse Events (participants affected / at risk) | 479/2507 | 451/2515
Other Adverse Events (participants affected / at risk) | 53/2507 | 60/2515
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rivaroxaban (N=2507) | Placebo (N=2515)
Anaemia (Blood and lymphatic system disorders) | 12 | 7
Anaemia Vitamin B12 Deficiency (Blood and lymphatic system disorders) | 1 | 0
Aplastic Anaemia (Blood and lymphatic system disorders) | 0 | 1
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 0 | 1
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 0 | 1
Cardiac Ventricular Thrombosis (Cardiac disorders) | 1 | 1
Cardiogenic Shock (Cardiac disorders) | 0 | 2
Cardiorenal Syndrome (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 1
Arteriovenous Malformation (Congenital, familial and genetic disorders) | 0 | 1
Buried Penis Syndrome (Congenital, familial and genetic disorders) | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 2
Vertigo Positional (Ear and labyrinth disorders) | 1 | 0
Basedow's Disease (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 1
Cataract (Eye disorders) | 7 | 2
Cataract Nuclear (Eye disorders) | 1 | 0
Diabetic Retinopathy (Eye disorders) | 1 | 0
Macular Hole (Eye disorders) | 1 | 0
Ophthalmoplegia (Eye disorders) | 0 | 1
Retinal Detachment (Eye disorders) | 1 | 0
Retinopathy Hypertensive (Eye disorders) | 0 | 1
Subretinal Fibrosis (Eye disorders) | 0 | 1
Visual Acuity Reduced (Eye disorders) | 1 | 0
Abdominal Adhesions (Gastrointestinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 6 | 7
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 1
Abdominal Tenderness (Gastrointestinal disorders) | 0 | 1
Anal Fissure (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Chronic Gastritis (Gastrointestinal disorders) | 3 | 1
Coeliac Disease (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 1
Dental Caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 2
Diverticulum Intestinal (Gastrointestinal disorders) | 1 | 0
Duodenal Obstruction (Gastrointestinal disorders) | 0 | 1
Duodenal Ulcer (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 3
Dysphagia (Gastrointestinal disorders) | 1 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Erosive Duodenitis (Gastrointestinal disorders) | 1 | 0
Food Poisoning (Gastrointestinal disorders) | 0 | 1
Gastric Ulcer (Gastrointestinal disorders) | 1 | 3
Gastritis (Gastrointestinal disorders) | 2 | 4
Gastritis Erosive (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Angiodysplasia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Necrosis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 3 | 1
Gastrooesophageal Sphincter Insufficiency (Gastrointestinal disorders) | 0 | 1
Hernial Eventration (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Ileus Paralytic (Gastrointestinal disorders) | 1 | 0
Incarcerated Inguinal Hernia (Gastrointestinal disorders) | 1 | 2
Incarcerated Umbilical Hernia (Gastrointestinal disorders) | 0 | 1
Inflammatory Bowel Disease (Gastrointestinal disorders) | 0 | 1
Inguinal Hernia (Gastrointestinal disorders) | 7 | 9
Intestinal Infarction (Gastrointestinal disorders) | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 5 | 0
Ischaemic Enteritis (Gastrointestinal disorders) | 0 | 1
Large Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Large Intestine Polyp (Gastrointestinal disorders) | 4 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Pancreatic Disorder (Gastrointestinal disorders) | 0 | 1
Pancreatic Necrosis (Gastrointestinal disorders) | 0 | 1
Pancreatitis Acute (Gastrointestinal disorders) | 3 | 3
Pancreatitis Chronic (Gastrointestinal disorders) | 2 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 0
Ulcerative Gastritis (Gastrointestinal disorders) | 1 | 0
Volvulus of Small Bowel (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 2
Asthenia (General disorders) | 5 | 1
Chest Discomfort (General disorders) | 0 | 1
Chest Pain (General disorders) | 0 | 1
Death (General disorders) | 0 | 3
Disuse Syndrome (General disorders) | 1 | 1
Drug Withdrawal Syndrome (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 2
General Physical Health Deterioration (General disorders) | 1 | 0
Heteroplasia (General disorders) | 0 | 1
Hyperthermia Malignant (General disorders) | 1 | 0
Impaired Healing (General disorders) | 1 | 1
Multiple Organ Dysfunction Syndrome (General disorders) | 5 | 3
Non-Cardiac Chest Pain (General disorders) | 7 | 6
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 4 | 4
Soft Tissue Inflammation (General disorders) | 1 | 0
Sudden Death (General disorders) | 1 | 0
Acute Hepatic Failure (Hepatobiliary disorders) | 1 | 0
Bile Duct Stone (Hepatobiliary disorders) | 0 | 1
Biliary Colic (Hepatobiliary disorders) | 1 | 0
Biliary Dilatation (Hepatobiliary disorders) | 1 | 0
Cardiac Cirrhosis (Hepatobiliary disorders) | 2 | 1
Cholangitis (Hepatobiliary disorders) | 3 | 1
Cholangitis Acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 10 | 5
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 7
Cholecystitis Chronic (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 3
Cirrhosis Alcoholic (Hepatobiliary disorders) | 1 | 0
Hepatic Cirrhosis (Hepatobiliary disorders) | 0 | 2
Hepatic Failure (Hepatobiliary disorders) | 2 | 1
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 | 1
Hepatic Lesion (Hepatobiliary disorders) | 0 | 1
Hepatitis Acute (Hepatobiliary disorders) | 1 | 0
Hepatorenal Failure (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 1
Liver Disorder (Hepatobiliary disorders) | 1 | 0
Portal Hypertension (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Sarcoidosis (Immune system disorders) | 1 | 0
Abdominal Abscess (Infections and infestations) | 1 | 0
Abscess (Infections and infestations) | 0 | 1
Abscess Limb (Infections and infestations) | 1 | 0
Abscess Soft Tissue (Infections and infestations) | 1 | 0
Anal Abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 3 | 1
Arthritis Bacterial (Infections and infestations) | 0 | 1
Bacterial Infection (Infections and infestations) | 0 | 1
Bacterial Sepsis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 12 | 9
Bronchitis Bacterial (Infections and infestations) | 1 | 0
Bursitis Infective (Infections and infestations) | 1 | 0
Carbuncle (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 7 | 7
Cellulitis Gangrenous (Infections and infestations) | 0 | 1
Cholecystitis Infective (Infections and infestations) | 2 | 0
Chronic Tonsillitis (Infections and infestations) | 1 | 0
Clostridium Difficile Colitis (Infections and infestations) | 1 | 1
Clostridium Difficile Infection (Infections and infestations) | 0 | 2
Cystitis (Infections and infestations) | 1 | 0
Dengue Fever (Infections and infestations) | 0 | 1
Device Related Infection (Infections and infestations) | 1 | 1
Diabetic Foot Infection (Infections and infestations) | 2 | 1
Diabetic Gangrene (Infections and infestations) | 1 | 3
Diverticulitis (Infections and infestations) | 0 | 1
Douglas' Abscess (Infections and infestations) | 0 | 1
Encephalitis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 2
Enteritis Infectious (Infections and infestations) | 0 | 1
Enterobacter Infection (Infections and infestations) | 0 | 1
Epididymitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 2 | 1
Escherichia Bacteraemia (Infections and infestations) | 1 | 0
Escherichia Infection (Infections and infestations) | 1 | 0
Escherichia Pyelonephritis (Infections and infestations) | 0 | 1
Escherichia Sepsis (Infections and infestations) | 0 | 3
Escherichia Urinary Tract Infection (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 7 | 4
Gastritis Viral (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 6 | 4
Gastroenteritis Shigella (Infections and infestations) | 0 | 1
Gastroenteritis Viral (Infections and infestations) | 1 | 0
Haemorrhagic Pneumonia (Infections and infestations) | 0 | 1
Hepatitis E (Infections and infestations) | 1 | 0
Herpes Zoster (Infections and infestations) | 0 | 1
Herpes Zoster Infection Neurological (Infections and infestations) | 0 | 1
Infected Dermal Cyst (Infections and infestations) | 1 | 0
Infected Skin Ulcer (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Infective Spondylitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 7 | 2
Intervertebral Discitis (Infections and infestations) | 1 | 0
Localised Infection (Infections and infestations) | 3 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 2 | 0
Lung Abscess (Infections and infestations) | 0 | 1
Lung Infection (Infections and infestations) | 8 | 6
Medical Device Site Infection (Infections and infestations) | 1 | 3
Meningitis (Infections and infestations) | 0 | 1
Myiasis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 4 | 1
Pancreas Infection (Infections and infestations) | 0 | 1
Parotid Abscess (Infections and infestations) | 0 | 1
Periodontitis (Infections and infestations) | 2 | 1
Peritonitis (Infections and infestations) | 5 | 3
Pharyngeal Abscess (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 68 | 72
Pneumonia Bacterial (Infections and infestations) | 1 | 5
Pneumonia Klebsiella (Infections and infestations) | 1 | 0
Pneumonia Staphylococcal (Infections and infestations) | 1 | 0
Post Procedural Infection (Infections and infestations) | 1 | 0
Postoperative Wound Infection (Infections and infestations) | 1 | 0
Pulmonary Tuberculosis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 2 | 0
Pyelonephritis Acute (Infections and infestations) | 0 | 3
Pyuria (Infections and infestations) | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 10 | 8
Sepsis (Infections and infestations) | 16 | 7
Septic Shock (Infections and infestations) | 4 | 6
Sinusitis (Infections and infestations) | 0 | 1
Staphylococcal Sepsis (Infections and infestations) | 1 | 0
Syphilis (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 1
Urinary Tract Infection (Infections and infestations) | 14 | 9
Urinary Tract Infection Bacterial (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0
Viral Myocarditis (Infections and infestations) | 0 | 1
Wound Infection (Infections and infestations) | 1 | 2
Accidental Overdose (Injury, poisoning and procedural complications) | 2 | 2
Alcohol Poisoning (Injury, poisoning and procedural complications) | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 1
Bone Fissure (Injury, poisoning and procedural complications) | 1 | 0
Burns Third Degree (Injury, poisoning and procedural complications) | 1 | 0
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 5 | 3
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 | 3
Femur Fracture (Injury, poisoning and procedural complications) | 8 | 4
Fibula Fracture (Injury, poisoning and procedural complications) | 0 | 1
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 1
Foreign Body (Injury, poisoning and procedural complications) | 1 | 0
Gun Shot Wound (Injury, poisoning and procedural complications) | 0 | 1
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 1
Head Injury (Injury, poisoning and procedural complications) | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 6 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 2
Intentional Overdose (Injury, poisoning and procedural complications) | 0 | 1
Limb Injury (Injury, poisoning and procedural complications) | 1 | 1
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1
Multiple Fractures (Injury, poisoning and procedural complications) | 2 | 1
Patella Fracture (Injury, poisoning and procedural complications) | 0 | 1
Pneumothorax Traumatic (Injury, poisoning and procedural complications) | 0 | 1
Post Procedural Complication (Injury, poisoning and procedural complications) | 1 | 0
Postoperative Renal Failure (Injury, poisoning and procedural complications) | 1 | 0
Postoperative Wound Complication (Injury, poisoning and procedural complications) | 2 | 0
Radiation Pneumonitis (Injury, poisoning and procedural complications) | 0 | 1
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 3 | 3
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 2 | 3
Tendon Rupture (Injury, poisoning and procedural complications) | 1 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 2 | 3
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 1
Ulna Fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Biopsy Pleura (Investigations) | 0 | 1
Biopsy Prostate (Investigations) | 1 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 1
Blood Creatinine Increased (Investigations) | 0 | 2
Blood Glucose Abnormal (Investigations) | 1 | 0
Blood Glucose Fluctuation (Investigations) | 0 | 1
Hepatic Enzyme Increased (Investigations) | 3 | 0
Liver Function Test Increased (Investigations) | 0 | 1
Oesophagogastroduodenoscopy (Investigations) | 0 | 1
Platelet Count Decreased (Investigations) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 1
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Diabetes Mellitus (Metabolism and nutrition disorders) | 7 | 8
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 9 | 3
Diabetic Ketosis (Metabolism and nutrition disorders) | 0 | 1
Diabetic Metabolic Decompensation (Metabolism and nutrition disorders) | 2 | 4
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0 | 1
Fluid Retention (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 3
Hyperglycaemic Hyperosmolar Nonketotic Syndrome (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 7
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 5 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 5
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Insulin-Requiring Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1
Lactic Acidosis (Metabolism and nutrition disorders) | 1 | 0
Metabolic Disorder (Metabolism and nutrition disorders) | 1 | 1
Type 1 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 5 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Foot Deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Gouty Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 4 | 1
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 4
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Polymyalgia Rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Spinal Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 3
Bladder Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Breast Cancer Stage Ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Clear Cell Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 3
Colon Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ear Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Epiglottic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gallbladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Gastric Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrooesophageal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic Cancer Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hypopharyngeal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intestinal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Lung Carcinoma Cell Type Unspecified Stage Ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 7
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant Neoplasm of Unknown Primary Site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Metastases to Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastatic Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Monoclonal Gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm of Orbit (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oropharyngeal Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Pancreatic Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Plasma Cell Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
Prostate Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate Cancer Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostatic Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal Cancer Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Renal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small Intestine Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Testis Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Throat Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tongue Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tongue Neoplasm Malignant Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amyotrophic Lateral Sclerosis (Nervous system disorders) | 1 | 0
Brain Injury (Nervous system disorders) | 1 | 0
Brain Oedema (Nervous system disorders) | 0 | 1
Carpal Tunnel Syndrome (Nervous system disorders) | 0 | 1
Cervicobrachial Syndrome (Nervous system disorders) | 0 | 1
Dementia (Nervous system disorders) | 2 | 0
Diabetic Neuropathy (Nervous system disorders) | 0 | 1
Dizziness Postural (Nervous system disorders) | 1 | 1
Encephalopathy (Nervous system disorders) | 1 | 1
Epilepsy (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 0 | 1
Hemianopia (Nervous system disorders) | 0 | 1
Hypoglycaemic Coma (Nervous system disorders) | 0 | 1
Hypoxic-Ischaemic Encephalopathy (Nervous system disorders) | 0 | 1
Intercostal Neuralgia (Nervous system disorders) | 0 | 1
Ischaemic Neuropathy (Nervous system disorders) | 0 | 1
Loss of Consciousness (Nervous system disorders) | 2 | 1
Lumbosacral Radiculopathy (Nervous system disorders) | 0 | 1
Metabolic Encephalopathy (Nervous system disorders) | 0 | 1
Neuroglycopenia (Nervous system disorders) | 0 | 1
Neuropathy Peripheral (Nervous system disorders) | 2 | 0
Sciatica (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 6 | 3
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1
Vertebrobasilar Insufficiency (Nervous system disorders) | 1 | 0
Device Dislocation (Product Issues) | 0 | 2
Alcohol Abuse (Psychiatric disorders) | 1 | 0
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 1 | 0
Alcoholism (Psychiatric disorders) | 1 | 0
Antisocial Personality Disorder (Psychiatric disorders) | 0 | 1
Anxiety Disorder (Psychiatric disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 2 | 1
Illness Anxiety Disorder (Psychiatric disorders) | 0 | 1
Major Depression (Psychiatric disorders) | 1 | 2
Psychotic Disorder Due to A General Medical Condition (Psychiatric disorders) | 0 | 1
Self-Injurious Ideation (Psychiatric disorders) | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 0 | 1
Suicide Attempt (Psychiatric disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 17 | 28
Calculus Urinary (Renal and urinary disorders) | 1 | 1
Chronic Kidney Disease (Renal and urinary disorders) | 14 | 7
Diabetic Nephropathy (Renal and urinary disorders) | 1 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
End Stage Renal Disease (Renal and urinary disorders) | 2 | 1
Glomerulonephritis (Renal and urinary disorders) | 1 | 0
Iga Nephropathy (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 3 | 0
Nephropathy Toxic (Renal and urinary disorders) | 1 | 0
Nephrotic Syndrome (Renal and urinary disorders) | 0 | 1
Prerenal Failure (Renal and urinary disorders) | 2 | 0
Renal Artery Stenosis (Renal and urinary disorders) | 1 | 0
Renal Colic (Renal and urinary disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 12 | 12
Renal Impairment (Renal and urinary disorders) | 4 | 9
Ureterolithiasis (Renal and urinary disorders) | 2 | 0
Urethral Stenosis (Renal and urinary disorders) | 1 | 0
Urinary Retention (Renal and urinary disorders) | 3 | 1
Urinary Tract Disorder (Renal and urinary disorders) | 1 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 4 | 1
Cystocele (Reproductive system and breast disorders) | 0 | 1
Gynaecomastia (Reproductive system and breast disorders) | 1 | 1
Ovarian Cyst Torsion (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Uterine Polyp (Reproductive system and breast disorders) | 0 | 1
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 15 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Dyspnoea Paroxysmal Nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Necrotising Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 9 | 5
Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vocal Cord Thickening (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 1
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetic Foot (Skin and subcutaneous tissue disorders) | 6 | 4
Dyshidrotic Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Hypersensitivity Vasculitis (Skin and subcutaneous tissue disorders) | 0 | 2
Necrobiosis Lipoidica Diabeticorum (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash Macular (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 2
Toxic Epidermal Necrolysis (Skin and subcutaneous tissue disorders) | 0 | 1
Anal Sphincterotomy (Surgical and medical procedures) | 1 | 0
Bile Duct Stent Removal (Surgical and medical procedures) | 0 | 1
Breast Tumour Excision (Surgical and medical procedures) | 1 | 0
Cataract Operation (Surgical and medical procedures) | 3 | 2
Chemotherapy (Surgical and medical procedures) | 0 | 1
Cyst Removal (Surgical and medical procedures) | 0 | 1
Debridement (Surgical and medical procedures) | 1 | 0
Diabetes Mellitus Management (Surgical and medical procedures) | 1 | 0
Drug Therapy (Surgical and medical procedures) | 0 | 1
Hernia Repair (Surgical and medical procedures) | 0 | 1
Ileostomy (Surgical and medical procedures) | 1 | 0
Inguinal Hernia Repair (Surgical and medical procedures) | 2 | 0
Insertion of Ambulatory Peritoneal Catheter (Surgical and medical procedures) | 1 | 0
Leg Amputation (Surgical and medical procedures) | 1 | 0
Peripheral Artery Bypass (Surgical and medical procedures) | 1 | 0
Prosthetic Vessel Implantation (Surgical and medical procedures) | 1 | 0
Removal of Ambulatory Peritoneal Catheter (Surgical and medical procedures) | 1 | 0
Spinal Fusion Surgery (Surgical and medical procedures) | 1 | 0
Spinal Laminectomy (Surgical and medical procedures) | 1 | 0
Transurethral Prostatectomy (Surgical and medical procedures) | 0 | 1
Aortic Aneurysm (Vascular disorders) | 1 | 0
Aortic Dissection (Vascular disorders) | 1 | 0
Arterial Haemorrhage (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1
Circulatory Collapse (Vascular disorders) | 2 | 1
Cryoglobulinaemia (Vascular disorders) | 0 | 1
Diabetic Vascular Disorder (Vascular disorders) | 0 | 1
Extremity Necrosis (Vascular disorders) | 3 | 0
Hypertension (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 4 | 2
Hypovolaemic Shock (Vascular disorders) | 2 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 2
Peripheral Arterial Occlusive Disease (Vascular disorders) | 0 | 1
Peripheral Ischaemia (Vascular disorders) | 2 | 0
Peripheral Vascular Disorder (Vascular disorders) | 1 | 0
Phlebitis Superficial (Vascular disorders) | 0 | 1
Subclavian Artery Stenosis (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rivaroxaban (N=2507) | Placebo (N=2515)
Nasopharyngitis (Infections and infestations) | 53 | 60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2016-12-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT01877915/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-12): https://cdn.clinicaltrials.gov/large-docs/15/NCT01877915/SAP_001.pdf